CLINICAL TRIAL: NCT04818645
Title: Insertable Cardiac Monitor for Primary Atrial Fibrillation Detection in High-Risk Heart Failure Patients (ASSERT-AF)
Brief Title: Insertable Cardiac Monitor for Primary Atrial Fibrillation Detection in High-Risk Heart Failure Patients
Acronym: ASSERT-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Ilan Goldenberg, Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00007311
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: Implantable cardiac monitor; Atrial fibrillation; Heart failure; Remote monitoring; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Stroke

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 fashion to undergo implant of an ASSERT ICM implant with remote monitoring and symptom-triggered mobile app transmissions versus conventional follow-up without an ICM. Randomization will be stratified by the degree of LV dysfunction to ensure balanced enrollment of HF subjects with mild LV dysfunction (LVEF = 36%-49%) and those with preserved LVEF (≥ 50% [i.e. heart failure with preserved ejection fraction - HFpEF]).
Who Masked: Outcomes Assessor
Masking Description: Events Review Committee: A blinded three-member Events Review Committee will review de-identified source documents obtained from each of the enrolling sites that will only be labelled with a subject ID. No data will be provided indicating the randomized treatment arm to the study and appropriately redacted with no ICM data provided. The information will be used to determine the nature of any clinical and adverse events. Available medical records and source documents will be used to determine cause-specific mortality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ASSERT insertable cardiac monitor (Experimental): The ASSERT implantable cardiac monitor (ICM) is an FDA-approved device that can be injected into the subcutaneous tissue and can provide automatic as well as patient triggered electrocardiographic recordings of symptomatic episodes during long term follow-up. This Implantable cardiac monitor is paired with a remote monitoring smartphone application called My Merlin that capable of rapid remote review of electrograms to be utilized in this study for arrhythmia detection. The ASSERT ICM is indicated for the monitoring and diagnostic evaluation of patients who experience unexplained symptoms such as: dizziness, palpitations, chest pain, syncope, and shortness of breath, as well as patients who are at risk for cardiac arrhythmias. It is also indicated for patients who have been previously diagnosed with atrial fibrillation or who are susceptible to developing atrial fibrillation.
  Interventions: Device: ASSERT Insertable Cardiac Monitor
- Conventional Management (Active Comparator): The conventional management arm will use arrhythmia signs and symptoms to determine occurrence of arrhythmias.
  Interventions: Other: Conventional Management and monitoring

INTERVENTIONS:
Device: ASSERT Insertable Cardiac Monitor — Subjects will be subcutaneously implanted with an Abbott ASSERT ICM with the device implant procedure per standard of care and current labelling. Data related to subjects' arrhythmias, via the Merlin.net Patient CareNetwork will be transmitted on a monthly basis to the treating physician and subsequently to the study coordination and database center (CCRC) at the University of Rochester. Data on the frequency/types of symptomatic (patient triggered) versus ICM detected (asymptomatic) arrhythmic events will be collected and adjudicated. Clinical data on medication, device interventions, cardiovascular events will be collected at follow-up visits.
  Arms: ASSERT insertable cardiac monitor
Other: Conventional Management and monitoring — Subjects randomized to the conventional management arm of the trial will undergo arrhythmia monitoring based on clinical indications and per standard available modalities including periodic electrocardiograms (ECG), Holter and/or event monitoring.
  Arms: Conventional Management

SUMMARY:
Patients with heart failure (HF) represent a large population of patients who are at high risk for complications related to undiagnosed atrial fibrillation (AF). However, currently there are limited modalities for early AF detection and subsequent stroke prevention in this high-risk population. An implantable cardiac monitor (ICM) is inserted subcutaneously and can provide long term arrhythmia information via remote monitoring.

The ASSERT-AF study seeks to accurately define the burden of AF and other arrhythmias in high-risk HF patients using an ASSERT ICM.

DETAILED DESCRIPTION:
Over 6 million people in the United States suffer from heart failure (HF). By the year 2030 the prevalence of HF is expected to exceed 8 million people. Heart failure accounts for 1 million hospital admissions each year, costing our economy in excess of $30 billion dollars per year. Mortality in patients with HF remains high, and nearly half of all patients diagnosed with HF will die within 5 years. More than half of all patients admitted with HF decompensation have preserved left ventricular systolic function. Patients with HF and mildly reduced or preserved left ventricular systolic function are at high risk for developing atrial fibrillation (AF), the occurrence of which often contributes to HF decompensation and increases morbidity and all-cause mortality. Similarly, patients with AF are at high risk for developing HF due to loss of atrio-ventricular synchrony and rapid uncontrolled ventricular rates. Detection of AF can be challenging and may go undiagnosed in asymptomatic or minimally symptomatic patients through conventional monitoring methods. Patients with HF represent a large population who are at risk for complications related to undiagnosed AF. AF increases the risk of stroke five-fold and the risk of death nearly two-fold. Moreover, strokes related to AF are twice as likely to be fatal or severely disabling compared to strokes due to other causes, such as ischemic small vessel disease or atheromatous large vessel disease. Cardiac implantable electronic devices (CIEDs), can be used for the early detection of AF in asymptomatic or mildly symptomatic patients with HF. However, current guidelines provide an indication for prophylactic implantable cardioverter defibrillator (ICD) only in HF patients with left ventricular ejection fraction (LVEF) ≤ 35%, whereas there are limited data for device-based detection of AF in HF patients with more preserved LVEF.

Implantable cardiac monitors (ICM) are devices that can be injected into the subcutaneous tissue and can provide automatic electrocardiographic recordings of asymptomatic arrhythmias as well as patient triggered electrocardiographic recordings of symptomatic episodes during long term follow-up. Implantable cardiac monitors are be paired with remote monitoring systems, capable of rapid remote review of electrograms. Accordingly, we hypothesize that a management strategy that incorporates ICM implantation in patients with HF and LVEF >35% will result in a significantly higher rate of AF detection leading to arrhythmia related interventions compared to conventional monitoring and follow-up in patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients more than 18 years of age (no upper age limit)
* HF exacerbation requiring initiation or augmentation of decongestive therapy in a hospital setting (hospitalization or emergency department visit) during the past 24 calendar months prior to consent date OR current treatment with loop-diuretics (furosemide, bumetanide, or torsemide).
* LVEF > 35% on a cardiac imaging study (echocardiogram, nuclear imaging, cardiac magnetic resonance imaging) performed during the past 24 calendar months prior to consent date
* One or more FDA-approved indications for an Abbott ICM (unexplained symptoms such as: dizziness, palpitations, chest pain, syncope, and shortness of breath, as well as patients who are at risk for cardiac arrhythmias).
* Willing to undergo an Abbott ICM implant and agree to remote ICM monitoring.

Exclusion Criteria:

* Existing implantable cardioverter defibrillator (ICD), biventricular ICD, implantable cardiac monitor or pacemaker.
* Known or documented history AF or atrial flutter any time in past.
* Has had a heart transplant
* Participation in other clinical trials (observational registries are allowed with approval from the Coordination Center)
* Unable or unwilling to cooperate with the protocol
* Unable or unwilling to sign the consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Median Time to first detection of AF lasting > 5 minutes | 24 months
  Defined as ICM detected AF in the intervention (implantable cardiac monitor) arm or captured by clinical symptoms and documented by ECG or Holter in the conventional arm.

SECONDARY OUTCOMES:
Time to initiation of guideline directed anti-arrhythmic and HF interventions | 24 months
  Interventions such AF ablation, initiation of antiarrhythmic, anticoagulation, beta-blocker therapy and others.
Number cardiovascular hospitalizations or death | 24 months
  Total number of cardiovascular hospitalizations or death in each arm.
Compare healthcare utilization using Abbott ICM vs. non-ICM monitoring. | 24 months
  Including emergency department visits, unplanned office visits, cardiovascular hospitalization or death
Mean quality of life measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 24 months
  All KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Mean percentage of time spent in atrial fibrillation (AF Burden) | 24 months
  AF burden, defined as average percentage of time spent in AF (i.e. amount of time spent in AF divided by the total amount of time a patient was monitored). AF burden will be quantified only in the intervention arm.
Time to detection of composite of arrhythmic events endpoint | 24 months
  Arrhythmic events consisting of AF, sustained ventricular tachycardia, and high-risk bradyarrhythmias (high degree AV block or sinus pause > 5 seconds), whichever occurs first.

OTHER OUTCOMES:
Compare the effect of patient-triggered transmissions on the time to Abbott ICM detection of arrhythmic events triggered by symptomatic recordings versus automatically detected arrhythmic event recordings. | 24 months
Evaluate the rate of actionable interventions following symptom triggered event versus the rate of actionable interventions associated with automatic detected arrhythmic events. | 24 months
  Including initiation of oral anticoagulation, guideline directed medical therapy, device and procedural interventions.
Correlate ICM interrogation data relating to heart sounds, body posture, activity, sleep detection and heart rate variability, with the risk of new heart failure events. | 24 months
  Such as hospitalizations, ED visits, unplanned office visits, out patients treatment with intravenous diuretic.

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Kannel WB, Wolf PA, Benjamin EJ, Levy D. Prevalence, incidence, prognosis, and predisposing conditions for atrial fibrillation: population-based estimates. Am J Cardiol. 1998 Oct 16;82(8A):2N-9N. doi: 10.1016/s0002-9149(98)00583-9. PMID 9809895
- [Background] Lin HJ, Wolf PA, Kelly-Hayes M, Beiser AS, Kase CS, Benjamin EJ, D'Agostino RB. Stroke severity in atrial fibrillation. The Framingham Study. Stroke. 1996 Oct;27(10):1760-4. doi: 10.1161/01.str.27.10.1760. PMID 8841325
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Lin HJ, Wolf PA, Benjamin EJ, Belanger AJ, D'Agostino RB. Newly diagnosed atrial fibrillation and acute stroke. The Framingham Study. Stroke. 1995 Sep;26(9):1527-30. doi: 10.1161/01.str.26.9.1527. PMID 7660392
- [Background] Anter E, Jessup M, Callans DJ. Atrial fibrillation and heart failure: treatment considerations for a dual epidemic. Circulation. 2009 May 12;119(18):2516-25. doi: 10.1161/CIRCULATIONAHA.108.821306. No abstract available. PMID 19433768
- [Background] Trulock KM, Narayan SM, Piccini JP. Rhythm control in heart failure patients with atrial fibrillation: contemporary challenges including the role of ablation. J Am Coll Cardiol. 2014 Aug 19;64(7):710-21. doi: 10.1016/j.jacc.2014.06.1169. PMID 25125304
- [Background] Maisel WH, Stevenson LW. Atrial fibrillation in heart failure: epidemiology, pathophysiology, and rationale for therapy. Am J Cardiol. 2003 Mar 20;91(6A):2D-8D. doi: 10.1016/s0002-9149(02)03373-8. PMID 12670636
- [Background] Pellicori P, Urbinati A, Kaur K, Zhang J, Shah P, Kazmi S, Capucci A, Cleland JGF, Clark AL. Prevalence and Incidence of Atrial Fibrillation in Ambulatory Patients With Heart Failure. Am J Cardiol. 2019 Nov 15;124(10):1554-1560. doi: 10.1016/j.amjcard.2019.08.018. Epub 2019 Aug 23. PMID 31558271
- [Background] Ducharme A, Swedberg K, Pfeffer MA, Cohen-Solal A, Granger CB, Maggioni AP, Michelson EL, McMurray JJ, Olsson L, Rouleau JL, Young JB, Olofsson B, Puu M, Yusuf S; CHARM Investigators. Prevention of atrial fibrillation in patients with symptomatic chronic heart failure by candesartan in the Candesartan in Heart failure: Assessment of Reduction in Mortality and morbidity (CHARM) program. Am Heart J. 2006 Jul;152(1):86-92. PMID 16838426
- [Background] Reiffel JA, Verma A, Kowey PR, Halperin JL, Gersh BJ, Wachter R, Pouliot E, Ziegler PD; REVEAL AF Investigators. Incidence of Previously Undiagnosed Atrial Fibrillation Using Insertable Cardiac Monitors in a High-Risk Population: The REVEAL AF Study. JAMA Cardiol. 2017 Oct 1;2(10):1120-1127. doi: 10.1001/jamacardio.2017.3180. PMID 28842973
- [Background] Beinart SC, Natale A, Verma A, Amin A, Kasner S, Diener HC, Pouliot E, Franco N, Mittal S. Real-World Use of Prophylactic Antibiotics in Insertable Cardiac Monitor Procedures. Pacing Clin Electrophysiol. 2016 Aug;39(8):837-42. doi: 10.1111/pace.12886. Epub 2016 Jun 7. PMID 27198480